CLINICAL TRIAL: NCT06212752
Title: A Phase 3 Randomized, Open-label Clinical Study to Evaluate the Pharmacokinetics and Safety of Subcutaneous Pembrolizumab Coformulated With Hyaluronidase (MK-3475A) Versus Intravenous Pembrolizumab, Administered With Chemotherapy, in the First-line Treatment of Participants With Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of Subcutaneous (SC) Pembrolizumab Coformulated With Berahyaluronidase Alfa (MK-3475A) vs Intravenous Pembrolizumab in Adult Participants With Metastatic Non-small Cell Lung Cancer (NSCLC) (MK-3475A-D77)-Japan Extension
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475A-D77 Japan Extension; MK-3475A-D77 (Other: MSD); 2022-501506-36-00 (Other: EU CT); jRCT2031230049 (Other: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Cisplatin; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy (Experimental): Japanese participants with treatment-naïve metastatic NSCLC receive 790 mg of Pembrolizumab Formulated with Berahyaluronidase Alfa via subcutaneous (SC) injection on Day 1 of each 6-week cycle for18 cycles (up to approximately108 weeks) in combination with platinum doublet chemotherapy.
  Interventions: Biological: Pembrolizumab (+) Berahyaluronidase alfa; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Filgrastim; Drug: Pegylated filgrastim
- Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy (Active Comparator): Japanese participants with treatment-naïve metastatic NSCLC receive 400 mg pembrolizumab intravenous (IV) infusion on Day 1 of each 6-week cycle for 18 cycles (up to approximately 108 weeks) in combination with platinum doublet chemotherapy.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Biological: Pembrolizumab; Drug: Filgrastim; Drug: Pegylated filgrastim

INTERVENTIONS:
Biological: Pembrolizumab (+) Berahyaluronidase alfa — Pembrolizumab (+) Berahyaluronidase alfa SC will be administered for squamous and nonsquamous NSCLC as per the schedule specified in arm; participants may be eligible for second course.
  Other Names: MK-3475A
  Arms: Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy
Drug: Pemetrexed — Pemetrexed 500 mg/m² by IV Infusion will be administered for nonsquamous NSCLC as per the schedule specified in arm.
  Other Names: Alimta
Drug: Cisplatin — Cisplatin 75 mg/m² by IV Infusion will be administered for nonsquamous and squamous NSCLC as per the schedule specified in arm.
  Other Names: Platinol-AQ
Drug: Carboplatin — Carboplatin AUC 5 mg/mL/min in nonsquamous and AUC 6 mg/mL/min in squamous NSCLC will be administered as per the schedule specified in arm.
Drug: Paclitaxel — Paclitaxel 200 mg/m² by IV Infusion will be administered for squamous NSCLC as per the schedule specified in arm.
  Other Names: Taxol
Drug: Nab-paclitaxel — Nab-paclitaxel 100 mg/m² by IV Infusion will be administered for squamous NSCLC as per the schedule specified in arm.
  Other Names: Albumin-bound paclitaxel
Biological: Pembrolizumab — Pembrolizumab by IV Infusion will be administered for squamous and nonsquamous NSCLC as per the schedule specified in arm; participants may be eligible for second course.
  Other Names: MK-3475, KEYTRUDA
  Arms: Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Drug: Filgrastim — Filgrastim will be administered as per the schedule specified for the arm.
Drug: Pegylated filgrastim — Pegylated filgrastim will be administered as per the schedule specified for the arm.

SUMMARY:
This study is to assess the pharmacokinetics (PK) and safety of SC pembrolizumab (+) berahyaluronidase alfa vs intravenous (IV) pembrolizumab, administered with chemotherapy in first line treatment of adult Japanese participants with metastatic non-small cell lung cancer. The primary hypotheses of this study are pembrolizumab (+) berahyaluronidase alfa subcutaneous (SC) is noninferior to pembrolizumab IV with respect to PK parameters.

DETAILED DESCRIPTION:
Japan extension study will require approximately six years which includes one additional year (beyond the global study's last participant last study related contact) from the time the first participant (or their legally acceptable representative) provides informed consent until the last participant's last study related contact to complete.

The Japan extension study will include participants previously enrolled in Japan in the global study for MK-3475A-D77 (NCT05722015) plus the study will continue to enroll participants in Japan until the sample size for participants in Japan reaches approximately 39.

As of Amendment 1 of the supplemental statistical analysis plan (effective date: 23 Aug 2024), patient reported outcomes will no longer be the secondary outcome measures of the study.

ELIGIBILITY:
The key inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has histologically or cytologically confirmed diagnosis of squamous or non-squamous Non-small Cell Lung Cancer (NSCLC)
* Must provide archival tumor tissue sample or newly obtained core, incisional, or excisional biopsy of a tumor lesion not previously irradiated
* Has a life expectancy of at least 3 months

Exclusion Criteria:

* Has a diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements
* Has received prior systemic anticancer therapy for metastatic NSCLC
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization
* Has received prior radiotherapy within 2 weeks of start of study intervention or has radiation-related toxicity requiring corticosteroids
* Has received radiation therapy to the lung (>30 Gray) within 6 months of start of study intervention
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has an active infection requiring systemic therapy
* Has a history of human immunodeficiency virus (HIV) infection
* Has a history of Hepatitis B or C
* Has not adequately recovered from major surgery or has ongoing surgical complications
* Has a history of allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2028-05-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (18):
- Japan (18):
  - Fujita Health University ( Site 4406), Toyoake, Aichi-ken
  - Kurume University Hospital ( Site 4412), Kurume, Fukuoka
  - Gunma Prefectural Cancer Center ( Site 4416), Otashi, Gunma
  - National Hospital Organization Hokkaido Cancer Center ( Site 4415), Sapporo, Hokkaido
  - Kanagawa Cardiovascular and Respiratory Center ( Site 4404), Yokohama, Kanagawa
  - Miyagi Cancer Center ( Site 4401), Natori-shi, Miyagi
  - Sendai Kousei Hospital ( Site 4400), Sendai, Miyagi
  - Kurashiki Central Hospital ( Site 4409), Kurashiki, Okayama-ken
  - Kansai Medical University Hospital ( Site 4408), Hirakata, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 4414), Takatsuki, Osaka
  - Saitama Prefectural Cancer Center ( Site 4402), Ina-machi, Saitama
  - Shizuoka Cancer Center ( Site 4405), Nagaizumi-cho,Sunto-gun, Shizuoka
  - Tochigi Cancer Center ( Site 4417), Utsunomiya, Tochigi
  - Juntendo University Hospital ( Site 4413), Bunkyo-ku, Tokyo
  - National Hospital Organization Kyushu Medical Center ( Site 4411), Fukuoka
  - National Hospital Organization Kyushu Cancer Center ( Site 4410), Fukuoka
  - Osaka International Cancer Institute ( Site 4407), Osaka
  - Nippon Medical School Hospital ( Site 4403), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 39 Japanese participants were randomized and received treatment (global study [NCT05722015; n=23] or to the extension portion [n=16]).
Groups:
- Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy: Japanese participants with treatment-naïve metastatic NSCLC receive 790 mg of Pembrolizumab Formulated With Berahyaluronidase Alfa via subcutaneous (SC) injection on Day 1 of each 6-week cycle for 18 cycles (up to approximately 108 weeks) in combination with platinum doublet chemotherapy.
Period: Overall Study
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Started | 28 | 11
Completed | 0 | 0
Not Completed | 28 | 11
Not completed — Death | 5 | 3
Not completed — Participants ongoing | 23 | 8

BASELINE CHARACTERISTICS:
Population: All Japanese participants who were randomized to the global study (NCT05722015) or to the extension portion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy | Total
Number analyzed (Participants) | 28 | 11 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (9.0) | 70.7 (8.2) | 69.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 24 | 8 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 11 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 28 | 11 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
  Participants
    ECOG = 0 | 18 | 6 | 24
    ECOG = 1 | 10 | 5 | 15
Histology (squamous vs. nonsquamous) [Count of Participants; unit: Participants] — Participants were classified according to tumor histology: Squamous or Non-squamous. The tumor histology determined potential treatment regimen.
  Participants
    Non-squamous | 14 | 9 | 23
    Squamous | 14 | 2 | 16
Programmed Cell Death Ligand 1 (PD-L1) Status [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Randomization of participants in the study was stratified by PD-L1 tumor proportion score (TPS) at baseline (<1%, 1-49%, ≥50% or Unknown). Higher percentages of PD-L1 TPS staining correspond to higher positivity of PD-L1 on a tumor.
  Participants
    TPS <1% | 12 | 6 | 18
    TPS 1-49% | 11 | 4 | 15
    TPS ≥50% | 2 | 1 | 3
    Unknown | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1) as assessed by blinded independent central review (BICR). The percentage of participants with CR or PR were reported.
Time Frame: Up to ~ 16 months
Population: All Japanese participants who were randomized to the global study (NCT05722015) or to the extension portion.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 28 | 11
Percentage of participants | 64.3 [44.1 to 81.4] | 18.2 [2.3 to 51.8]

2. Secondary Outcome: Cycle 1: Area Under the Curve From Time 0 to 6 Weeks (AUC0-6 Weeks) of Pembrolizumab After the First Dose
Description: AUC0-6 weeks was defined as a measure of pembrolizumab exposure that was calculated as the product of serum drug concentration and time from zero to 6 weeks. Blood samples were collected at pre-specified timepoints to determine AUC0-6 weeks. Per protocol, geometric mean AUC0-6 weeks value of pembrolizumab after the first dose of pembrolizumab formulated with berahyaluronidase alfa in arm 1 and after first dose of pembrolizumab in arm 2 was presented.
Time Frame: Cycle 1: Arm 1: Day 1: Predose and Days 2, 3, 4, 5, 6, 7, 10, 15, 29, and 42 postdose; Arm 2: Day 1: Predose and at the end of infusion, Days4, 15, 29, and 42 postdose (cycle length = 42 days)
Population: All Japanese participants who were randomized to the global study (NCT05722015) or to the extension portion who received a dose in Cycle 1 with at least 1 valid postdose pharmacokinetic (PK) sample available in Cycle1 and for whom a model-based assessment of AUC0-6 weeks could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg·day/mL
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 28 | 11
µg·day/mL | 1864.76 (22.18) | 1697.98 (18.50)
Statistical Analysis 1: Comparison: Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy vs Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy; Test type: Non-Inferiority — Non-inferiority margin is 0.8; Geometric Mean Ratio (GMR) = 1.10, 95% CI 2-sided [0.95 to 1.27] — GMR and associated 96% confidence interval (Cl) were calculated using the Welch's t test. GMR was calculated as geometric mean (GM) of Pembrolizumab Formulated with Berahyaluronidase Alfa to GM of Pembrolizumab

3. Secondary Outcome: Cycle 3: Trough Serum Concentration (Ctrough) of Pembrolizumab at Steady State
Description: Ctrough is defined as the trough concentration at steady-state. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Ctrough.
Time Frame: Cycle 3: Arm 1: Day 1: Predose and Days 4, 10, and 42 postdose; Arm 2: Day 1: Predose and at the end of infusion, Days 4 and 42 postdose (cycle length = 42 days)
Population: All Japanese participants who were randomized to the global study (NCT05722015) or to the extension portion who received a dose in Cycle 1 and Cycle 3 with at least 1 valid postdose PK sample available in Cycle 1through Cycle 3 and for whom a model-based assessment of Ctrough could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/ml
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 24 | 7
µg/ml | 45.11 (35.58) | 30.86 (24.93)
Statistical Analysis 1: Comparison: Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy vs Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy; Test type: Non-Inferiority — Non-inferiority margin is 0.8; GMR = 1.46, 95% CI 2-sided [1.14 to 1.88] — GMR and associated 95% CI were calculated using the Welch's t test. GMR was calculated as geometric mean (GM) of Pembrolizumab Formulated with Berahyaluronidase Alfa to GM of Pembrolizumab

4. Secondary Outcome: Cycle 1: Maximum Serum Concentration (Cmax) of Pembrolizumab After the First Dose
Description: Cmax was defined as the maximum serum concentration of pembrolizumab reached after first dose. Blood samples were collected at pre-specified timepoints for the determination of Cmax. Per protocol, geometric mean Cmax value of pembrolizumab after the first dose of pembrolizumab formulated with berahyaluronidase alfa in arm 1 and after first dose of pembrolizumab in arm 2 was presented.
Time Frame: Cycle 1: Arm 1: Day 1: Predose and Days 2, 3, 4, 5, 6, 7, 10, 15, 29, and 42 postdose; Arm 2: Day 1: Predose and at the end of infusion, Days 4, 15, 29, and 42 postdose (cycle length = 42 days)
Population: All Japanese participants who were randomized to the global study (NCT05722015) or to the extension portion who received who received a dose in Cycle 1 with at least 1 valid postdose PK sample available in Cycle 1 and for whom a model-based assessment of Cmax could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/ml
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 28 | 11
µg/ml | 71.54 (23.7) | 141.9 (16.4)

5. Secondary Outcome: Cycle 1: Trough Serum Concentration (Ctrough) of Pembrolizumab After the First Dose
Description: Ctrough was defined as the lowest serum concentration of pembrolizumab reached after first dose. Blood samples were collected at pre-specified timepoints for the determination of Ctrough. Per protocol, geometric mean Ctrough value of pembrolizumab after the first dose of pembrolizumab formulated with berahyaluronidase alfa in arm 1 and after first dose of pembrolizumab in arm 2 was presented.
Time Frame: At designated time points (Up to ~28 months)
Population: All Japanese participants who were randomized to the global study (NCT05722015) or to the extension portion who received a dose in Cycle 1 with at least 1 valid postdose PK sample available in Cycle 1 and for whom a model-based assessment of Ctrough could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/ml
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 28 | 11
µg/ml | 23.62 (27.9) | 16.27 (29.7)

6. Secondary Outcome: Cycle 3: Area Under the Curve From Time 0 to 6 Weeks (AUC0-6 Weeks) of Pembrolizumab at Steady State
Description: AUC0-6 weeks was defined as a measure of pembrolizumab exposure that was calculated as the product of serum drug concentration and time from zero to 6 weeks. Blood samples were collected at pre-specified timepoints to determine AUC0-6 weeks. Per protocol, geometric mean AUC0-6 weeks value of pembrolizumab at steady state of pembrolizumab formulated with berahyaluronidase alfa in arm 1 and pembrolizumab in arm 2 was presented.
Time Frame: At designated time points (Up to ~28 months)
Population: All Japanese participants who were randomized to the global study (NCT05722015) or to the extension portion who received a dose in Cycle 1 and Cycle 3 with at least 1 valid postdose PK sample available in Cycle 1 through Cycle 3 and for whom a model-based assessment of AUC0-6 weeks could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•day/ml
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 24 | 7
µg•day/ml | 3116 (27.3) | 2514 (17.3)

7. Secondary Outcome: Cycle 3: Maximum Serum Concentration (Cmax) of Pembrolizumab at Steady State
Description: Cmax was defined as the maximum serum concentration of pembrolizumab reached at steady state. Blood samples were collected at pre-specified timepoints to determine Cmax. Per protocol, geometric mean Cmax value of pembrolizumab at steady state of pembrolizumab formulated with berahyaluronidase alfa in arm 1 and pembrolizumab in arm 2 was presented.
Time Frame: as for outcome 3
Population: All Japanese participants who were randomized to the global study (NCT05722015) or to the extension portion who received a dose in Cycle 1 and Cycle 3 with at least 1 valid postdose PK sample available in Cycle 1 through Cycle 3 and for whom a model-based assessment of Cmax could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 24 | 7
µg/mL | 108.1 (25.3) | 159.8 (13.2)

8. Secondary Outcome: Number of Participants Who Test Positive for Anti-Drug Antibodies (ADAs) for Pembrolizumab
Description: Blood samples are to be collected at designated time points for the determination of the presence or absence of anti-pembrolizumab antibodies. The percentage of participants who develop anti pembrolizumab antibodies will be reported.
Time Frame: At designated time points (Up to ~28 months)
Reporting Status: Not Posted

9. Secondary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 by BICR or death due to any cause, whichever occurs first.
Time Frame: Up to ~59 months
Reporting Status: Not Posted

10. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause.
Time Frame: Up to ~59 months
Reporting Status: Not Posted

11. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1)
Description: For participants who show confirmed CR or PR, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Time Frame: Up to ~59 months
Reporting Status: Not Posted

12. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with an AE will be reported for Arms 1 and 2.
Time Frame: Up to~28 months
Reporting Status: Not Posted

13. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported for Arms 1 and 2.
Time Frame: Up to~25 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to approximately 16 months
Description: All-Cause Mortality includes all randomized Japanese participants. Serious & Other adverse events (AEs) include all randomized Japanese participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer was not considered an AE unless considered related to study treatment. MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment were excluded as AEs. Data were reported by treatment received.
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
All-Cause Mortality (participants affected / at risk) | 5/28 | 3/11
Serious Adverse Events (participants affected / at risk) | 12/28 | 3/11
Other Adverse Events (participants affected / at risk) | 28/28 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy (N=28) | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy (N=28) | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy (N=11)
Anaemia (Blood and lymphatic system disorders) | 12 (12) | 9 (12)
Leukopenia (Blood and lymphatic system disorders) | 6 (17) | 3 (5)
Neutropenia (Blood and lymphatic system disorders) | 13 (32) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (16) | 4 (8)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 5 (5) | 1 (1)
Epiretinal membrane (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Punctate keratitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 11 (12) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (15) | 3 (7)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (3) | 1 (3)
Malaise (General disorders) | 3 (5) | 2 (6)
Oedema (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 3 (4) | 2 (2)
Pyrexia (General disorders) | 6 (6) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 5 (7) | 4 (7)
Amylase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 3 (5)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (4)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 3 (3) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (2)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (4)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (3)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 4 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (5)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (3)
Headache (Nervous system disorders) | 1 (3) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Any information identified by the Sponsor as confidential must be deleted prior to submission.

DOCUMENTS (2):
  • Study Protocol (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT06212752/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT06212752/SAP_001.pdf